CLINICAL TRIAL: NCT03950180
Title: Assessing The Impact Of Incorporating Charlson Comorbidity Scores On Patient Anxiety And Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benaroya Research Institute (Other)
Collaborators: Virginia Mason Hospital/Medical Center (Other); Axio Research Corporation (Industry)
Responsible Party: Principal Investigator, John Corman, MD, Principal Investigator, Benaroya Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB13054
Record Dates: First submitted 2019-05-09; First posted 2019-05-15 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCCI group (Active Comparator): In addition to standard of care counseling the additional provision of the patient's specific Prostate Cancer Comorbidity Index score and life expectancy estimation was provided.
  Interventions: Other: Prostate Cancer Comorbidity Index (PCCI) score
- Standard care (No Intervention): Standard of care was defined as prostate cancer counseling reflecting the best practices of a multidisciplinary team of urologists, radiation oncologists and medical oncologists.

INTERVENTIONS:
Other: Prostate Cancer Comorbidity Index (PCCI) score — Life expectancy information
  Arms: PCCI group

SUMMARY:
The purpose of this study was to determine whether providing patients with life expectancy (LE) information in the form of their Prostate Cancer Comorbidity Index (PCCI) scores impacted their decisional conflict or anxiety about prostate cancer or death.

DETAILED DESCRIPTION:
Patients with newly diagnosed prostate cancer were consented and randomized to receive standard of care counseling (SOC) versus the same counseling plus provision of their specific LE (PCCI). Patients were blinded to the specific content of their counseling session. After counseling, patients completed the Decisional Conflict Scale (DCS), Death Anxiety Scale (DAS), Memorial Anxiety Scale for Prostate Cancer (MAX-PC), and Patient Satisfaction Questionnaire (PSQ-18). Treatment preferences were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Men 18 years and older
* Newly diagnosed prostate cancer

Exclusion Criteria:

* Non-English speaking
* Prior history of prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 277 (Actual)
Dates: Start 2013-07-12 (Actual); Primary Completion 2015-02-27 (Actual); Study Completion 2015-02-27 (Actual)

PRIMARY OUTCOMES:
Traditional Decisional Conflict Scale (DCS) | within 120 days of receiving counseling
  This is to assess the ability to implement decisions. Each of the 16 questions range from strongly agree (a score of 1), to strongly disagree (a score of 5). The total score could be as low as 16 or as high as 80. A lower total score represents a better outcome, with a score of <25 associated with the ability to implement decisions and a score of >37.5 associated with decision delay and feeling unsure.

SECONDARY OUTCOMES:
The Modified 18-item Memorial Anxiety Scale for Prostate Cancer | within 120 days of receiving counseling
  This is to assess anxiety about prostate cancer. Each of the 18 questions range from not at all (a score of 1) to often (a score of 4). The total score could range from 18 to 72. A lower total score indicates less anxiety about prostate cancer and a lower score represents the better the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: John M Corman, MD, Principal Investigator — Benaroya Research Institute at Virginia Mason

IPD SHARING:
Plan to Share IPD: No